CLINICAL TRIAL: NCT06810544
Title: A Phase 1/2, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, and Preliminary Antitumor Activity of TNG456 Monotherapy and in Combination With Abemaciclib in Patients With Solid Tumors With MTAP Loss
Brief Title: Safety and Tolerability of TNG456 Alone and in Combination With Abemaciclib in Patients With Solid Tumors With MTAP Loss
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tango Therapeutics, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNG456-C101
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; Glioma Glioblastoma Multiforme; Glioma, Malignant; Solid Tumor; Non-Small Cell Adenocarcinoma; Lung Cancer; Brain Tumor
Keywords: MTAP; PRMT5 inhibitor; CDK 4/6; abemaciclib; Tango
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Glioblastoma; Glioma; Lung Neoplasms; Brain Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation (sequential) followed by phase 2 dose expansion (parallel)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Single Agent and Combination Dose Escalation (Experimental): Solid tumor participants with confirmed MTAP loss will receive escalating doses of TNG456 single agent and in combination with abemaciclib to estimate the MTD
  Interventions: Drug: TNG456; Drug: abemaciclib
- NSCLC Single Agent Dose Expansion (Experimental): NSCLC (squamous and non squamous) participants with confirmed MTAP loss will receive TNG456 at the identified RP2D(s)
  Interventions: Drug: TNG456
- GBM Single Agent Dose Expansion (Experimental): GBM participants with confirmed MTAP loss will receive TNG456 at the identified RP2D(s)
  Interventions: Drug: TNG456
- Tumor Agnostic Single Agent Dose Expansion (Experimental): Patients with specific solid tumor types that have a confirmed MTAP loss will receive TNG456 at the identified RP2D(s)
  Interventions: Drug: TNG456
- NSCLC Combination Expansion (Experimental): NSCLC (squamous and non-squamous) participants with confirmed MTAP loss will receive TNG456 at the identified RP2D(s) with abemaciclib
  Interventions: Drug: TNG456; Drug: abemaciclib
- GBM Combination Expansion (Experimental): GBM participants with confirmed MTAP loss will receive TNG456 at the identified RP2D(s) with abemaciclib
  Interventions: Drug: TNG456; Drug: abemaciclib
- Tumor Agnostic Combination Expansion (Experimental): Participants with specific tumor types with confirmed MTAP loss will receive TNG456 at the identified RP2D(s) with abemaciclib
  Interventions: Drug: TNG456; Drug: abemaciclib

INTERVENTIONS:
Drug: TNG456 — A selective PRMT5 inhibitor
Drug: abemaciclib — A kinase inhibitor
  Other Names: Verzenio
  Arms: GBM Combination Expansion; NSCLC Combination Expansion; Single Agent and Combination Dose Escalation; Tumor Agnostic Combination Expansion

SUMMARY:
This is a first in human study of TNG456 alone and in combination with abemaciclib in patients with advanced or metastatic solid tumors known to have an MTAP loss. The first part of the study is an open-label, dose escalation and the second part is an open label dose expansion in specific solid tumor types with a confirmed MTAP loss. The study drug, TNG456, is a selective PRMT5 inhibitor administered orally. The study is planned to treat up to 191 participants.

DETAILED DESCRIPTION:
This is a Phase 1/2 multi-center, open label study in solid tumor patients who have a confirmed MTAP loss in their tumor. The Phase 1 portion is a dose escalation study of oral TNG456 administered as a single agent and in combination with oral abemaciclib in solid tumor patients with confirmed MTAP loss. In the Phase 2 expansion part of the study, 6 arms defined by confirmed tumor types will enroll in parallel at the RP2D(s) of TNG456 and in combination. In both parts of the study participants who tolerate the drug may continue treatment until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Has a tumor with a confirmed MTAP loss
* Is ≥18 years of age at the time of signature of the main study ICF
* Has had progression or an inadequate response to or is intolerant of the approved standard of care therapy, no standard of care therapy exists, or the investigator has determined that treatment with the standard of care therapy is not appropriate.
* Is able to swallow tablets
* Adequate Organ function/reserve per local labs
* Negative serum pregnancy test result at screening
* Has an ECOG performance status score of 0 to 1
* Has measurable disease based on RECIST v1.1 or a confirmed glioblastoma (IDH-wildtype) with radiographic evidence of disease progression or recurrence defined by RANO 2.0.
* Has an ECOG performance score of 0 to 1 or for GBM has a Karnofsky performance status score ≥70.

Exclusion Criteria:

* A female patient is who is pregnant or breastfeeding
* Has impaired GI function or disease that may significantly alter the absorption of oral study treatment(s)
* Has an active infection requiring systemic therapy
* Has received prior treatment with a PRMT5 inhibitor or a MAT2A inhibitor
* Patients in the expansion receiving the combination therapy that have received prior treatment with a CDK4/6 inhibitor
* Clinically relevant cardiovascular disease
* Has a prior or ongoing clinically significant illness may affect the safety of the patient, impair the assessment of study results or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Maximum Tolerated Dose | 21 days
  To determine the MTD, recommended dose(s) (RD), and dosing schedule of TNG456 monotherapy and in combination with abemaciclib
Phase 2 Anti-neoplastic Activity Single Agent | 18 weeks
  To assess the antitumor activity of TNG456 in patients with advanced or metastatic solid tumors with MTAP loss by RECIST or modified RANO criteria
Phase 2 Anti-neoplastic Activity Combination Treatment | 18 weeks
  To assess the antitumor activity of TNG456 in combination with abemaciclib in patients with advanced or metastatic tumors with MTAP loss by RECIST or modified RANO criteria

SECONDARY OUTCOMES:
Phase 1 Anti-neoplastic Activity Single Agent | 18 weeks
  To assess preliminary evidence of antitumor activity of TNG456 in patients with advanced solid tumors with MTAP loss by RECIST or modified RANO criteria
Phase 1 and 2 Adverse Event Profile | 21 days
  To describe the safety and tolerability profile of TNG456 as a monotherapy and in combination with abemaciclib
Phase 1 and 2 Concentration versus Time Curve | 16 days
  Measure the area under the plasma concentration versus time curve (AUC)
Phase 1 and 2 Time to Achieve Maximal Plasma Concentration | 16 days
  Measure the time to achieve maximal plasma concentration (Tmax)
Phase 1 and 2 Maximum Observed Plasma Concentration | 16 days
  Measure the maximum observed plasma concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Tab Cooney, MD, Study Director — Tango Therapeutics, Inc.
Locations (13):
- United States (13):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of California, Irvine, Irvine, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No